CLINICAL TRIAL: NCT03881280
Title: The System Fammeal Comprising an App With Tailored Recommendations and Gamification for Parents to Counteract Childhood Obesity, at Health Care Centers - Pilot Randomized Control Trial
Brief Title: The System Fammeal With Tailored Recommendations and Gamification for Parents to Counteract Childhood Obesity
Acronym: Fammeal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Administração Regional de Saúde do Norte, Portugal (Other); Agrupamento de Centros de Saúde do Grande Porto III - Maia / Valongo, Portugal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FCT-PD/BD/128309/2017
Record Dates: First submitted 2019-03-12; First posted 2019-03-19 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2019-08

CONDITIONS: Overweight and Obesity
Keywords: Childhood Obesity; Nutrition; mHealth; Parenting
MeSH Terms: conditions — Overweight; Obesity; Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Treatment as usual for 4 weeks
- Intervention group (Experimental): Education through the app for 4 weeks
  Interventions: Behavioral: Parenting education program

INTERVENTIONS:
Behavioral: Parenting education program — Parenting education program through the app Fammeal. It includes educational content, tailored to parents and centered on positive parenting child-feeding practices. The app will also include a virtual-pet game for children, in order to help them self-regulate their intake.
  Through the app, parents will:
  * Fill in a registration questionnaire, which will tailor recommendations.
  * Receive information and video content recommendations.
  * Set goals related to their child's lifestyle and tracking progress.
  * Earn points by watching the contents.
  * Invite children to play a serious game.
  * Exchange messages with other users.
  The investigators created a support website that connects to the main server to get data gathered from the mobile app and game.
  Arms: Intervention group

SUMMARY:
The investigators aim to test an evidence-based intervention, allocated to a mobile app designed to parents and their children with 3 to 6 years old, identified by family doctors or nurses at well-child care visits as overweight or obese for age.

This intervention aims to improve parent's perceptions and attitudes regarding children's weight status and food intake, leading to better dietary intake and children's' eating behaviors through positive parental child-feeding practices. In this study, the investigators aim to assess the feasibility of the intervention and explore its impact on the beliefs and attitudes of parents.

DETAILED DESCRIPTION:
The investigators will enroll parents and their children with 3 to 6 years old, identified by family doctors or nurses at well-child care visits as overweight/obese for age.

Participant's eligibility will be assessed. Participants will be randomized to: 1) control group; 2) intervention group. The control group will receive treatment as usual. Parents in the intervention group will be provided with the app and invited to use it for 4 weeks. During the 4 weeks, the administrator monitors the app usage and call once to parents to improve it, if needed.

Both groups will perform a pre- and post-test, evaluating parent's perceptions and attitudes regarding children's weight status and food intake; eating behaviors and parental child-feeding practices.

ELIGIBILITY:
Inclusion Criteria:

* Children with 36 to 83 months at the start of the intervention.
* Children overweight or obese for age, according to World Health Organization criteria.
* Parent/ caregiver with at least 18 years old.
* Parent/caregiver involved in child feeding management (≥ 5 in a 0-10 rating scale, from 'Not at all' to 'Extremely involved').
* Parent/ caregiver able to read, speak and understand Portuguese.
* Parent/caregiver with an android device.
* Parent/caregiver willing to participate in the research study, to participate in two face-to-face evaluations, to install and use the app and to receive weekly notifications and 1-3 calls, during 4 weeks.

Exclusion Criteria:

* Children with any medical conditions that affect growth, intake or physical activity.
* Children with any dietary professional advice, in the last 6 months.

Ages: 36 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Perceptions and Attitudes regarding children's weight status at 4 weeks | Baseline and 4 weeks
  Parents recognize their children as overweight/obese (0-10 rating scale, ranging from 'too slim' to 'too heavy') and are concerned about it (0-10 rating scale, from 'Not concerned at all' to 'Extremely concerned').
Change from Baseline Perceptions and Attitudes regarding children's food intake at 4 weeks | Baseline and 4 weeks
  Parents are aware of dietary recommendations for children's age (Fruit and vegetables, sugar-sweetened beverages, energy-dense foods and water) and are concerned about their achievement (0-10 rating scale, from 'Not concerned at all' to 'extremely concerned').
Dietary Intake (in this pilot RCT only evaluated to test the randomization) | Baseline
  Increase fruit and vegetables and water intake per day and decrease sugar-sweetened beverages and energy-dense foods intake per week (evaluated by food frequency questionnaire).
Parental child-feeding practices (in this pilot RCT only evaluated to test the randomization) | Baseline
  Increase Availability and Accessibility of Healthy Foods; Attractive presentation of foods; Nutrition Education and decrease of Distractions (evaluated by HomeSTEAD Survey, adapted to Portuguese within this study).
Study population eligibility and interest | Baseline
  Proportion of all parents invited who meet eligibility and who accepted to enroll.
Participant engagement | 4 weeks
  Mean of points earned and app access per participant during intervention and proportion of recommended videos watched.

SECONDARY OUTCOMES:
Eating Behaviors (in this pilot RCT only evaluated to test the randomization). | Baseline
  Increase Children's Satiety Responsiveness. This was evaluated by the mean score of 5 items of Children's Eating Behavior Questionnaire.Satiety Responsiveness reflects the ability to regulate the amount of food eaten, based on perceived fullness. Parents answered in a 5-point Likert scale (0 = never; 5 = always), with higher values reflecting higher punctuation in each subscale. A version of this questionnaire has been previously validated and adapted to Portuguese children aged 3-13 years (Viana, Sinde, & Saxton, 2008).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Afonso, Principal Investigator — Faculdade de Psicologia e de Ciências da Educação da Universidade do Porto
Locations (1):
- Faculdade de Psicologia e de Ciências da Educação da Universidade do Porto, Porto, Porto, Portugal, Portugal

REFERENCES:
- [Result] Afonso L, Rodrigues R, Reis E, Miller KM, Castro J, Parente N, Teixeira C, Fraga A, Torres S. Fammeal: a gamified mobile application for parents and children to help health care centers treat childhood obesity. IEEE Transactions on Games. 2020. doi: 10.1109/TG.2020.3015804.
- [Result] Afonso L, Rodrigues R, Castro J, Parente N, Teixeira C, Fraga A, Torres S. A Mobile-Based Tailored Recommendation System for Parents of Children with Overweight or Obesity: A New Tool for Health Care Centers. Eur J Investig Health Psychol Educ. 2020 Aug 7;10(3):779-794. doi: 10.3390/ejihpe10030057. PMID 34542511
- See also: Website of the project — https://fammeal.up.pt/